CLINICAL TRIAL: NCT02451904
Title: Microvascular and Metabolic Dysregulation in the Pathogenesis of Severe and Cerebral Malaria Investigated Through Host Metabolomics
Brief Title: Severe and Cerebral Malaria Investigated Through Host Metabolomics
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Chittagong Medical College and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BAKMAL1407
Record Dates: First submitted 2015-05-15; First posted 2015-05-22 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Severe Malaria
Keywords: Pathogenesis; Microvascular function; Metabolic dysregulation; Metabolomics
MeSH Terms: conditions — Malaria | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, CSF, Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Severe/Cerebral Malaria: Intensive monitoring
  Interventions: Other: Observation
- Uncomplicated Malaria: Intensive monitoring
  Interventions: Other: Observation
- Sepsis: Intensive monitoring
  Interventions: Other: Observation
- Acidosis: Intensive monitoring
  Interventions: Other: Observation
- Encephalitis: Intensive monitoring
  Interventions: Other: Observation
- Healthy Individuals: Monitoring
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
* The aim is to describe disease mechanisms of severe and cerebral malaria and identify new targets for adjunctive therapies.
* Despite treatment between 10-30% of patients with severe malaria die.
* Metabolic acidosis and cerebral malaria are major complications associated with mortality across all age groups. Still, their underlying pathogenesis remains incompletely understood.
* Using a metabolomics approach, this study aims to characterise the spectrum of acids accumulating during acidosis, and investigate patterns of metabolic dysregulation associated with coma and seizures.

ELIGIBILITY:
Severe/Cerebral Malaria:

* Any P. falciparum parasitaemia detected by asexual stages on a peripheral blood-slide or a positive rapid diagnostic test in combination with one or more Modified WHO Criteria for Severe Malaria (Hien et al, 1996)
* < 24 hours after treatment commencement with either parenteral artemisinin or quinine
* Age > 12 years
* Full informed written consent obtained

Uncomplicated malaria:

* Any level of Plasmodium parasitaemia, detected by asexual stages on a peripheral blood-slide or a positive rapid diagnostic test without any of the complications of severe malaria stated above.
* Age > 12 years
* Full informed written consent obtained

Sepsis:

* Clinical signs of infection in combination with any two of the following signs:

  1. Heart rate > 90 beats per minute;
  2. Respiratory rate > 20 breaths per minute, a PaCO2 of < 32 mmHg, or the use of mechanical ventilation for an acute respiratory process;
  3. Tympanic temperature > 38°C or < 36 °C;
  4. White-cell count of > 12x109/L or < 4x109/L, or a differential count showing 10% immature neutrophils ;
* Negative peripheral blood slide for any stages of malaria parasites or a negative rapid diagnostic test for falciparum and vivax malaria
* [As bacterial culture is not routinely available at the study site, positivity of cultures is not required]
* Age > 12 years
* Full informed written consent obtained

Acidosis:

* Clinical suspicion of metabolic acidosis in combination with any of the following:

  1. Peripheral venous bicarbonate < 15 mmol/L
  2. Peripheral venous base excess < -3 mmol/L
* Negative peripheral blood slide for any stages of malaria parasites or a negative rapid diagnostic test for falciparum and vivax malaria; and not meeting any of the inclusion criteria for sepsis as stated above.
* Age > 12 years
* Full informed written consent obtained

Encephalitis:

* GCS < 11/15
* Documented fever > 38°C
* Onset of symptoms < 2 weeks, with an indication a lumbar puncture as part of the diagnostic work up
* Negative peripheral blood slide for any stages of malaria parasites or a negative rapid diagnostic test for falciparum and vivax malaria
* Age > 12 years
* Full informed written consent obtained

Healthy volunteers:

* No chronic or acute disease
* No fever in the past 2 weeks
* Age > 16 years
* Full informed written consent obtained

Exclusion Criteria:

* Known pre-existing chronic medical conditions including advanced hepatic disease.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In total, up to 840 patients may be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Characterisation of patterns of metabolic dysregulation in severe malaria | 4-6 weeks
  Interrelationship between disturbances in metabolic pathways associated with acidosis and cerebral malaria

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Arjen M. Dondorp, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Chittagong Medical College Hospital (CMCH), Chittagong, Bangladesh

REFERENCES:
- [Background] Dondorp A, Nosten F, Stepniewska K, Day N, White N; South East Asian Quinine Artesunate Malaria Trial (SEAQUAMAT) group. Artesunate versus quinine for treatment of severe falciparum malaria: a randomised trial. Lancet. 2005 Aug 27-Sep 2;366(9487):717-25. doi: 10.1016/S0140-6736(05)67176-0. PMID 16125588
- [Background] Dondorp AM, Fanello CI, Hendriksen IC, Gomes E, Seni A, Chhaganlal KD, Bojang K, Olaosebikan R, Anunobi N, Maitland K, Kivaya E, Agbenyega T, Nguah SB, Evans J, Gesase S, Kahabuka C, Mtove G, Nadjm B, Deen J, Mwanga-Amumpaire J, Nansumba M, Karema C, Umulisa N, Uwimana A, Mokuolu OA, Adedoyin OT, Johnson WB, Tshefu AK, Onyamboko MA, Sakulthaew T, Ngum WP, Silamut K, Stepniewska K, Woodrow CJ, Bethell D, Wills B, Oneko M, Peto TE, von Seidlein L, Day NP, White NJ; AQUAMAT group. Artesunate versus quinine in the treatment of severe falciparum malaria in African children (AQUAMAT): an open-label, randomised trial. Lancet. 2010 Nov 13;376(9753):1647-57. doi: 10.1016/S0140-6736(10)61924-1. Epub 2010 Nov 7. PMID 21062666
- [Derived] Leopold SJ, Ghose A, Allman EL, Kingston HWF, Hossain A, Dutta AK, Plewes K, Chotivanich K, Day NPJ, Tarning J, Winterberg M, White NJ, Llinas M, Dondorp AM. Identifying the Components of Acidosis in Patients With Severe Plasmodium falciparum Malaria Using Metabolomics. J Infect Dis. 2019 May 5;219(11):1766-1776. doi: 10.1093/infdis/jiy727. PMID 30566600